CLINICAL TRIAL: NCT00907530
Title: Phase IV, Double-Blind, Multi-Center, Randomized, Crossover Study to Compare 0.1 mmol/kg OF MULTIHANCE® WITH 0.1 mmol/kg OF GADOVIST® in Magnetic Resonance Imaging (MRI) of the Brain
Brief Title: Study to Compare MultiHance With Gadovist in Magnetic Resonance Imaging (MRI) of the Brain
Acronym: MERIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: MH-123
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Brain Lesions
MeSH Terms: interventions — gadobenic acid; gadobutrol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MULTIHANCE (Active Comparator): gadobenate dimeglumine
  Interventions: Drug: MULTIHANCE:
- GADOVIST (Active Comparator): gadobutrol
  Interventions: Drug: GADOVIST

INTERVENTIONS:
Drug: MULTIHANCE: — MULTIHANCE ® 0.5 M,0.1 mmol/kg
  Arms: MULTIHANCE
Drug: GADOVIST — GADOVIST ® 1.0 M,0.1 mmol/kg
  Arms: GADOVIST

SUMMARY:
This study is being conducted as a phase IV, double-blind, multi-center, randomized, crossover trial aimed at a within-subject comparison of MULTIHANCE and GADOVIST at a dose of 0.1 mmol/kg, in terms of qualitative and quantitative assessment of unenhanced MRI (UE MRI) and contrast-enhanced MRI (CE MRI) for the visualization of brain disease.

ELIGIBILITY:
Inclusion Criteria:

* Enroll subjects in this study if they meet the following inclusion criteria:
* Are at least 18 years of age or older
* Are able to give written informed consent and are willing to comply with the protocol requirements
* Are scheduled to undergo MRI
* Are willing to undergo two MRI procedures within 14 days
* Have confirmed or are highly suspected to have brain tumor(s) (primary or secondary), as determined by:
* clinical/neurological symptomatology;
* diagnostic testing, such as CT or previous MRI examinations; or
* have had recent surgery within 6 months and are to be evaluated for recurrence.

Exclusion Criteria:

* Exclude subjects from this study if they do not fulfill the inclusion criteria, or if any of the following conditions are observed.
* Are pregnant or lactating females. Exclude the possibility of pregnancy:
* by testing on site at the institution (serum or urine bHCG) within 24 h prior to the start of each investigational product administration
* by history (i.e., tubal ligation or hysterectomy)
* post menopausal with a minimum of 1 year without menses
* Have any known allergy to one or more of the ingredients in the investigational product, or have a history of hypersensitivity to any metals
* Have congestive heart failure (class IV according to the classification of the New York Heart Association
* Have suffered a stroke within a year
* Have received or are scheduled to receive any other contrast medium in the 24 h preceding through the 24 h following Exam 1, and in the 24 h preceding through the 24 h following Exam 2
* Have received or are scheduled to receive an investigational compound and/or medical device within 30 days before admission into the present study, through the 24 h post-administration of the second investigational product.
* Have moderate-to-severe renal impairment, defined as a GFR/eGFR < 60 mL/min.
* Have been previously entered into this study
* Have received or are scheduled for one of the following:
* Surgery within three weeks prior to the first examination or between the two examinations
* Initiation of steroid therapy between the two examinations
* Radiosurgery between the two examinations
* Have any contraindications to MRI such as a pace-maker, magnetic material (i.e., surgical clips) or any other conditions that would preclude proximity to a strong magnetic field.
* Are suffering from severe claustrophobia
* Have any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To show superiority of a 0.1 mmol/kg dose of MULTIHANCE as compared to 0.1 mmol/kg dose of GADOVIST, in terms of the by-subject global diagnostic preference between exams (i.e., based on predose + postdose image sets). | Day 1 and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Pirovano, MD, Study Director — Bracco Diagnostics
Locations (1):
- Hamilton Health Sciences Corporation, Hamilton, Ontario, Canada